CLINICAL TRIAL: NCT06514092
Title: Study on the Long-Term Risk of Recurrence of Anoperineal Fistula After Treatment with Anti-tumor Necrosis Factor (TNF) and Seton Drainage in Crohn's Disease : LT-SAFCD
Brief Title: Study on the Long-Term Risk of Recurrence of Anoperineal Fistula in Crohn's Disease
Acronym: LT-SAFCD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0174
Record Dates: First submitted 2024-07-11; First posted 2024-07-23 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Crohn Disease
Keywords: perianal fistula; anti-TNF; seton drainage; inflammatory bowel disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Crohn's patients
  Interventions: Other: anti-TNF therapy and seton drainage

INTERVENTIONS:
Other: anti-TNF therapy and seton drainage — Crohn's disease patients who have undergone treatment with anti-TNF therapy and seton drainage.

SUMMARY:
This research aims to evaluate the long-term recurrence risk of perianal fistulas in Crohn's disease patients who have undergone treatment with anti-TNF therapy and seton drainage.The research seeks to identify factors influencing recurrence and assess the long term effectiveness of these treatments in preventing fistula recurrence. This study will provide insights that could enhance treatment strategies and improve patient outcomes.

DETAILED DESCRIPTION:
Scientific Justification :

● Perianal fistulas are a common and challenging complication of Crohn's disease, significantly impacting patient quality of life. Infliximab, an TNFα antagonist has shown its efficacy in inducing remission of these fistulas. Seton drainage is often used alongside anti-TNF therapy to promote fistula healing and prevent abscess formation. However, data with long term follow up are still lacking on the impact of these treatments. Understanding the long-term outcomes of these combined treatments is crucial for optimizing therapeutic strategies and improving patient management.

Treatment Strategy :

● The treatment involves administering infliximab to control inflammation and promote fistula closure, along with seton drainage to maintain fistula patency and prevent abscesses, ensuring continuous drainage and reducing infection risk.

Follow-up Description :

● Patients are monitored retrospectively through medical records for a period ranging from several months to years, assessing recurrence rates and potential predictors of recurrence. Follow-up includes regular clinical evaluations, biological evaluations (blood test and fecal calprotectin), colonoscopy, imaging studies such as MRI, and patient-reported outcomes to gather comprehensive data on the long-term efficacy and safety of the combined treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Crohn's disease
* drainage of an anal fistula with seton combined with the initiation of anti-TNF alpha treatment
* Patient who was treated in the digestive center of the Toulouse University Hospital for drainage of an anal fistula between January 1, 2000 and December 31, 2010

Exclusion Criteria:

Patient followed less than 6 months after seton drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with crohn's disease
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Long-term recurrence-free survival rate of perianal fistulas | through study completion, an average of 2 years
  To evaluate the long-term recurrence-free survival rate of perianal fistulas after combined treatment with anti-TNF alpha and seton drainage

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LE COSQUER, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France